CLINICAL TRIAL: NCT04457180
Title: A Single Arm, Open and Fixed Sequence Study to Investigate the Pharmacokinetic Effects of Apatinib Mesylate on CYP2C8 Substrate Repaglinide or CYP2B6 Substrate in Advanced Solid Tumor Subjects
Brief Title: A Pharmacokinetic Interaction Study Between Apatinib Mesylate and Repaglinide or Bupropion in Advanced Solid Tumor Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-APTN-I-008
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — apatinib; repaglinide; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): In phase A, subjects receiving a single dose of Repaglinide orally on day 1 , a single dose of Bupropion orally on day 2 and wash-out for 10 days, then apatinib once daily will be conducted on D5 through D16
  # In addition, In phase B, subjects receiving a single dose of Repaglinide (in combination with apatinib) orally on day 12 , a single dose of Bupropion (in combination with apatinib) orally on day 13.
  Interventions: Drug: Apatinib Mesylate; Drug: Repaglinide; Drug: Bupropion

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib will be administered daily from on D5 through D16
Drug: Repaglinide — Repaglinide will be administered daily on D1 and D12
Drug: Bupropion — Bupropion will be administered daily on D2 and D13

SUMMARY:
The primary objective of the study was to assess investigate the pharmacokinetic effects of Apatinib Mesylate on CYP2C8 Substrate Repaglinide or CYP2B6 Substrate Bupropion and metabolite Hydroxy bupropion in Advanced solid tumor subjects.

The secondary objective of the study was to assess the safety of Apatinib or/and Repaglinide and Bupropion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old (Include both values).
2. Patients with histopathologically or cytologically confirmed advanced solid tumor (not necessary to have measurable lesions).
3. Refractory or intolerant to standard treatment regimens, or no effective standard treatment regimens available, or the patients refused to use standard treatment plan.
4. ECOG PS score: 0-1.
5. Expected survival ≥ 3 months.
6. Subjects have recovered from other treatments, at least 6 weeks since the last use of nitrosourea or mitomycin; at least 4 weeks since the last use of small molecule targeted therapy; at least 8 weeks since the last use of biological macromolecular therapy; at least 4 weeks since radiotherapy or surgery; at least 4 weeks since the last use of other cytotoxic or cytostatic drugs.
7. Major organs must function normally, meeting the following criteria: (1) Hematology (no blood transfusion or blood products within the last 14 days, not corrected with G-CSF or other hematopoietic colony-stimulating factors):

   a. HB≥100 g/L; b. ANC≥1.5×109/L; c. PLT≥90×109/L; (2) Blood biochemistry: d. TBIL≤ 1.25×ULN; e. ALT and AST≤2.5×ULN; f. ALP≤2.5×ULN; g. Serum Cr ≤ 1.5 × ULN or endogenous CrCl > 60 mL/min (Cockcroft-Gault formula); h. Albumin > 30 g/L.
8. Sign the ICF voluntarily, have good compliance, corporate with follow-up visits, and follow the study requirements.

Exclusion Criteria:

1. Gastric cancer; tumors with risk of bleeding which researchers evaluated.
2. Active brain metastasis (medically uncontrolled);
3. Symptomatic third space fluid that cannot be controlled by drainage or other methods;
4. Dysphagia, chronic diarrhea, or other factors affecting drug intake and absorption;
5. Uncontrolled hypertension;
6. Heart rate < 60, Grade II or greater myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (QTc interval ≥ 450 ms in males and ≥ 470 ms in females);
7. Contraindications to Repaglinide and Bupropion;
8. NYHA Class III-IV cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% by echocardiography;
9. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 s or APTT > 1.5 ULN), bleeding tendency or who are currently receiving thrombolytics;
10. Arterial/venous thrombosis within 6 months prior to the first dose;
11. Hemorrhage and thrombophilia;
12. Major surgery or with severe traumatic injury, fracture, or ulcer within 4 weeks prior to the first dose;
13. Abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months prior to the first dose;
14. Urine protein ≥ ++ and 24 h urine protein ≥ 1.0 g as indicated by urinalysis;
15. Treatment with steroids for more than 50 days, or requires chronic steroid use;
16. Use of study drugs in other clinical trials within 4 weeks prior to the first dose;
17. Use of drugs affected gastric acid secretion or inhibitors of cytochrome enzyme CYP2C8、CYP2B6、CYP2D6、CYP3A or transporter OATP1B1, or traditional Chinese medicine within 2 weeks prior to the first dose; use of inducers of metabolic enzymes CYP2C8, CYP2B6, CYP2D6, or CYP3A within 4 weeks prior to the first dose;
18. Unable to hold drugs that may prolong QT interval during the study (such as antiarrhythmics);
19. Habitual alcohol consumption or smoking, tested positive for alcohol screening, and unable to abstain from smoking and alcohol during the trial;
20. Other factors affecting drug absorption, distribution, metabolism, excretion within 48 hours；
21. Active hepatitis B (positive HBsAg and HBV-DNA≥104 or 2000IU/ml) or C (Hepatitis C antibodies are positive and HCV-RNA is above the detection limit of the analytical method);
22. Active infection requiring antimicrobial therapies (such as antibacterials, antivirals, or antifungals);
23. Immunodeficiency, including positive results of HIV test or other acquired or congenital immunodeficiencies, or a history of organ transplantation;
24. Allergic constitution, or known allergies to drug components used in this study;
25. Pregnant or lactating women;
26. Other factors that may affect the progress or the conclusion of the study, as determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of digoxin | through study completion, an average of 16 days
  Peak Plasma Concentration (Cmax) of digoxin
Pharmacokinetics parameter: AUC of digoxin | through study completion, an average of 16 days
  Area under the plasma concentration versus time curve (AUC) of digoxin

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of digoxin | through study completion, an average of 16 days
  Time of maximum observed concentration (Tmax) of digoxin
Pharmacokinetics parameter: T1/2 of digoxin | through study completion, an average of 16 days
  Half time (T1/2) of digoxin
Pharmacokinetic parameters CL/F of digoxin | through study completion, an average of 16 days
  Total body clearance for extravascular administration (CL/F) of digoxin
Pharmacokinetics parameter: Vz/F of digoxin | through study completion, an average of 16 days
  Volume of distribution (Vz/F) of digoxin
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 16 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant criteria

CONTACTS AND LOCATIONS:
Overall Officials: pan yueyin, Ph.D., Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided